CLINICAL TRIAL: NCT01921010
Title: Benefit of Elevation of HDL-cholesterol/Triglyceride Lowering on Cardiovascular Outcomes in Women
Brief Title: Benefit of Elevation of HDL-C in Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Noel Bairey Merz, Director, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3954
Record Dates: First submitted 2013-08-09; First posted 2013-08-13 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Cardiovascular Outcomes
MeSH Terms: interventions — Niacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Niaspan (Active Comparator): Patients will be randomized to Niaspan 1.5 g/d in addition to usual care statin lipid lowering agents. The dose of Niaspan will be titrated over a 4-week period and then patients will remain on study drug for additional 12 weeks. The dose of statin will be adjusted in a blinded fashion in both groups at week 10 to similarly achieve a LDL-C of less than 100mg/dl.
  Interventions: Drug: Niaspan
- Control (Placebo Comparator): patients will be randomized to placebo 1.5 g/d in addition to usual care statin lipid lowering agents. The dose of placebo will be titrated over a 4-week period and then patients will remain on study drug for additional 12 weeks. The dose of statin will be adjusted in a blinded fashion in both groups at week 10 to similarly achieve a LDL-C of less than 100mg/dl.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Niaspan — See Arm Description
  Arms: Niaspan
Drug: Placebo — See Arm Description
  Arms: Control

SUMMARY:
The combination of HDL-C elevation, lowering of triglycerides and further LDL-C reduction accomplished by the addition of niacin to statin medication would improve endothelial function as compared to LDL-C reduction alone in patients with and without coronary artery disease and the combination of low HDL-C/high triglycerides.

The combination of lipid lowering therapy would have beneficial effects on markers of inflammation. These benefits would be particularly evident in women.

ELIGIBILITY:
Inclusion Criteria:

* Stable CAD(coronary artery disease) patients on statin therapy with LDL-C between 90-135mg/dl and triglycerides > 150mg/dl
* Well-controlled diabetes with HbA1C < 7.5 currently on statin therapy, able to tolerate Niacin without unstable blood glucose levels with LDL-C between 90-135mg/dl and triglycerides > 150mg/dl
* Stable patients on statin therapy with LDL-C between 90-135mg/dl and triglycerides > 150mg/dl

Exclusion Criteria:

* History of MI(myocardial infarction), PTCA(percutaneous transluminal coronary angiography) or surgery within previous 3 months
* Currently on Niaspan and unwilling to withdraw Niaspan therapy or known intolerance to niacin
* Active or known gall bladder disease
* Pregnant or nursing women
* Significant comorbidity that precludes participation
* Significant liver disease, active alcoholism, or LFT(liver function test) >1.5x's ULN( upper limit of normal) at screening
* Diabetes with Hg A1C(hemoglobin A1c) < 7.5
* PI perceived inability to comply with protocol

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2003-06; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
endothelial function | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: C. Noel Bairey Merz, M.D., Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes